CLINICAL TRIAL: NCT00816413
Title: T Cell-Reduced Unrelated Donor Allogeneic Peripheral Blood Stem Cell Transplantation With Pentostatin and Low-Dose Total Body Irradiation
Brief Title: Donor Stem Cell Transplant, Pentostatin, and Total-Body Irradiation in Treating Patients With Hematological Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Screenings yielded inadequate eligible subjects to enroll.
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0164-07-FB; P30CA036727 (NIH)
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Nonmalignant Neoplasm
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; essential thrombocythemia; polycythemia vera; primary myelofibrosis; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; marginal zone B-cell lymphoma of mucosal lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; aplastic anemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; contiguous st II adult diffuse small cleaved cell lymphoma; noncontig stage II adult diffuse small cleaved cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neoplasms; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Anemia, Aplastic; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclosporine; Cyclosporins; Mycophenolic Acid; Pentostatin; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Flow Cytometry; Immunoenzyme Techniques; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Donor Stem Cell Transplant, Pentostatin & Total-Body Irradiation for Hematological Cancer (Experimental): This phase I/II trial is studying the side effects of giving a donor stem cell transplant after pentostatin and total-body irradiation and to see how well it works in treating patients with hematological cancer.
  Interventions: Drug: cyclosporine; Drug: mycophenolate mofetil; Drug: pentostatin; Genetic: cytogenetic analysis; Genetic: fluorescence in situ hybridization; Genetic: protein analysis; Other: flow cytometry; Other: immunoenzyme technique; Other: laboratory biomarker analysis; Other: reduced-intensity transplant conditioning procedure; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation (PBSC); Radiation: total-body irradiation

INTERVENTIONS:
Drug: cyclosporine — 2 mg/kg IV over 2 hours every 12 hours starting at 0700 on days -1, 0, and +1 (total of six doses).
  Other Names: Gengraf, Neoral, and Sandimmune
Drug: mycophenolate mofetil — 15 mg/kg orally twice a day starting day 0 until day +27 then stopped without tapering in the absence of aGVHD then tapered over two months in the absence of aGVHD. Doses will be rounded to the nearest 250 mg.
  Other Names: CellCept
Drug: pentostatin — 4 mg/m2/d IV over 30 minutes daily x 3 days, (days -10, -9, -8)to begin ten days prior to stem cell infusion (Day 0).
  Other Names: Nipent
Genetic: cytogenetic analysis — At days +28 and +70 post-transplant, patients' blood will be evaluated for CD3 and overall WBC chimerism.
Genetic: fluorescence in situ hybridization — Mixed chimerism is defined as the detection of 95% or less donor T cells (CD3+), expressed as a proportion of the total T cell and WBC population as measured by DNA.
Genetic: protein analysis — Blood samples will be at baseline(day -11 or before) , days -8 and -1, prior to transplant on day 0, then weekly (days +7, +14, +21 and +28) post-transplant through day +28. Five ml's of blood will be drawn at each collection through a central line using heparinized vaccutainers. Samples will be spun down at 1200 g and plasma aspirated and stored in -80 oC until analyzed for the ELISA Assays being done for research purposes in this protocol.
Other: flow cytometry — Peripheral blood Peripheral blood flow cytometry for immunophenotyping including Th/c1 and Th/c2 subsets, mitogens (PHA, PWM), NK and LAK function studies, DCs, apoptosis assay of tumor cells, and lymphocyte subsets (CD4, CD8, CD19, CD56
Other: immunoenzyme technique — Peripheral blood for immunophenotyping including Th/c1 and Th/c2 subsets, mitogens (PHA, PWM), NK and LAK function studies, DCs, apoptosis assay of tumor cells, and lymphocyte subsets (CD4, CD8, CD19, CD56
Other: laboratory biomarker analysis — Donor mononuclear cells from the stem cell product (SCP) obtained with apheresis will be analyzed for surface markers, including CD3, CD4, CD8, CD19, CD14, CD56, TCR+CD8+ cells, Th/c1 and Th/c2, Fas and FasL, and DCs, as well as for apoptosis
Other: reduced-intensity transplant conditioning procedure — Allopurinol 300 mg orally once daily x 10 days, to begin one day prior to treatment with Pentostatin (day -11 to day -2) .
  Pentostatin 4 mg/m2/d IV over 30 minutes daily x 3 days, (days -10, -9, -8)to begin ten days prior to stem cell infusion (Day 0) .
  Pre and Post Pentostatin Hydration: 1000ml Normal Saline IV over 2 hours pre each dose of Pentostatin and 1000ml Normal Saline IV over 4 hours post each dose of Pentostatin on days -10, -9, -8.
  Pre Pentostatin Recommended Antiemetics: Ondansetron 32 mg IV over 30 minutes to be given 30 min. before each dose of Pentostatin on days -10, -9, -8. Alternative ondansetron equivalent or other ancillary antiemetics may be used at the discretion of the treating physician.
  Pred Forte Eye Drops: two drops in each eye every 4 hours while awake x 7 days after starting Pentostatin (day -10 to day -4).
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Each patient will receive up to four IV infusions administered over 30 minutes of donor T cells at increasing cell doses given at intervals.
Procedure: peripheral blood stem cell transplantation (PBSC) — PBSC are infused intravenously either by infusion or IV push on day 0 through a secure intravenous access (i.e. the double-lumen central catheter place pre transplant) according to institutional guidelines.
Radiation: total-body irradiation — 2.0 GY will be administered on day -1. Total-body irradiation (TBI) will consist of 2.0 GY at 8-12cGy/min via 6MV photons delivered AP/PA fields, without lung blocks or via lateral fields with lucite compensator along the head and neck region. TLD (thermal luminescent dosimetry) will be used to verify dose uniformity. It is anticipated that TBI will be given on day -1; however, the timing of TBI administration may be altered by factors beyond the control of the Principal Investigator because of the delivery of unrelated donor stem cells.

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Removing the T cells from the donor cells before transplant and giving cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase I/II trial is studying the side effects of giving a donor stem cell transplant after pentostatin and total-body irradiation and to see how well it works in treating patients with hematological cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety of pentostatin and low-dose total body irradiation followed by T-cell-reduced unrelated donor peripheral blood stem cell transplantation, in terms of regimen-related toxicity, in patients with hematological malignancies.
* To evaluate the efficacy of this regimen, measured as engraftment rate and establishment of donor hematopoietic chimerism, in these patients.

Secondary

* To determine the incidence of acute and chronic graft-versus-host disease in patients treated with this regimen.

OUTLINE:

* Reduced-intensity preparative regimen: Patients receive pentostatin IV over 30 minutes once daily on days -10 to -8 and undergo low-dose total-body irradiation on day -1.
* Unrelated donor peripheral blood stem cell transplantation (PBSCT): Patients undergo T-cell-reduced donor PBSCT on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 2 hours twice daily on days -1, 0, and 1 and then orally twice daily on days 2-70 followed by a taper in the absence of GVHD. Patients also receive oral mycophenolate mofetil twice daily on days 0-27 followed by a taper.

Patients undergo bone marrow aspirate and biopsies and blood sample collection periodically for laboratory studies. Samples are analyzed for cytokines (i.e., IL-6, TNF-γ, IL-1β, and IL-10) by ELISA; phenotypic, molecular, and functional analysis of immunologic reconstitution markers (i.e., PHA, IL-2, IL-4, IL-10, IL-12, Fas, FasL, TNF, TGF-β, and IFN-γ) by flow cytometry; and cytogenetics by FISH.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria • Diagnosis of a confirmed hematological malignancy that has relapsed or is at high risk for relapsing, including any of the following:

Acute myeloid leukemia (AML) meeting any of the following criteria:

Antecedent hematologic disorder Therapy related Primary induction failure

In first complete remission (CR1) with poor-risk cytogenetics, as defined by the following:

del(5q)/-5 del(7q)/-7 abn(3q) t(6;9) del(20q) del(17p)

+13 Complex karyotype t(9;22) = 11q23 rearrangement In second complete remission (CR2) or greater

Acute lymphoblastic leukemia meeting any of the following criteria:

In CR1 with WBC > 50,000/mm³ at diagnosis

In CR1 with poor-risk cytogenetics (i.e., t[9;22], t[1;19], t[4;11]) AND meets at least 1 of the following criteria:

19-75 years of age AND received prior high-dose chemotherapy, total-body irradiation (TBI), or a radiation dose that precludes administration of 12 Gy of TBI = 50-75 years of age = 19-75 years of age with hematopoietic stem cell transplantation (HSCT) comorbidity index ≥ 3 CNS or testicular involvement at diagnosis No CR within 4 weeks of initial treatment Primary induction failure In CR2 or greater

Myelodysplastic syndromes meeting the following criteria:

Intermediate-2 or high-risk category as determined by International Prognostic Scoring System Not considered a candidate for intensive or standard chemotherapy or HSCT

Chronic myelogenous leukemia meeting any of the following criteria:

First chronic phase AND < 40 years of age First chronic phase AND no hematologic response after 3 months of imatinib mesylate therapy First chronic phase AND never achieved a complete cytogenetic response during imatinib mesylate therapy First chronic phase AND loss of previously documented response Accelerated phase Blast crisis phase Chronic myeloproliferative disorder (i.e., polycythemia vera, essential thrombocythemia, myelofibrosis) Bone marrow blasts > 5% and/or other evidence of progression to acute leukemia Chronic myelomonocytic leukemia Severe aplastic anemia Failed prior antithymocyte globulin and cyclosporine immunosuppressive therapy

Mantle cell lymphoma meeting any of the following criteria:

In CR1 In first partial remission (PR1) In CR2 or greater In second PR (PR2) or greater

Indolent non-Hodgkin lymphoma OR chronic lymphocytic leukemia meeting either of the following criteria:

In CR2 or greater In PR2 or greater Lymphoblastic lymphoma In CR1 or greater

Must have minimal residual disease as defined by either of the following:

No more than 5% blasts in blood and/or bone marrow (in patients with acute leukemia/MDS) No bulky adenopathy (> 5 cm masses) and/or < 20% bone marrow involvement by lymphoma (in patients with lymphoma) No progressive disease within 8 weeks of most recent prior therapy OR within 12 weeks of prior autologous HSCT No active CNS malignancy (i.e., known positive CSF cytology or parenchymal lesions visible by CT scan or MRI) HLA-matched unrelated peripheral blood stem cell donor available Meets the University of Nebraska Medical Center's or the National Marrow Donor Program's criteria for donors Matched at 7/8 or 8/8 HLA-A, B, C, or DRβ1 loci by molecular typing If match is not at allele level, suitability for donation requires discussion with and approval by the principal investigator Not an identical twin Karnofsky performance status 60-100% Creatinine clearance ≥ 55 mL/min Total bilirubin ≤ 2 times upper limit of normal (ULN) (unless due to Gilbert's disease or malignancy) ALT and AST ≤ 4 times ULN DLCO ≥ 40% FEV1/FVC ratio ≥ 50% of predicted Cardiac ejection fraction ≥ 40%Prior cytoreductive chemotherapy or irradiation to areas of bulky disease allowed, as determined by the primary physician in consultation with the study investigators

Exclusion Criteria No CR within 4 weeks of initial treatment No other concurrent anti-tumor therapy Not pregnant or nursing (fertile patients must use effective contraception) Not receiving supplementary continuous oxygen No NYHA grade II-IV cardiac disease HIV positive Active hepatitis B (i.e., positive HBsAg and/or positive HBeAg or high copy number on quantitative RNA testing) or hepatitis C Active uncontrolled infection or immediate life-threatening condition Uncontrolled medical illnesses (e.g., uncontrolled systemic hypertension or diabetes)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Severe transplant-related toxicity | before day 100
  Severe transplant-related toxicity (grade III-IV adverse events) as assessed by NCI CTCAE v2.0
Stable donor engraftment | by day 70
  Stable donor engraftment
Mortality | at day 100
  Death

SECONDARY OUTCOMES:
Incidence of grade III-IV acute graft-versus-host disease | at day 100
  An interim analysis will be performed after the accrual of each five patients (i.e., three interim analyses and 1 final analysis) has reached day 100.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bociek, MD, Principal Investigator — University of Nebraska